CLINICAL TRIAL: NCT04274530
Title: Cognitive Behavioral Therapy to Optimize Post-Operative Recovery (COPE): A Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy to Optimize Post-Operative Recovery Trial
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Orthopaedic Trauma Association (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COPE-Definitive
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Fractures, Closed; Fractures, Open
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Fractures, Closed; Fractures, Open | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants with operatively managed extremity fractures 2-12 weeks post-fracture fixation will be randomized to receive either cognitive behavioural therapy (CBT) delivered through a mobile application or standard of care (control). Outcomes will be assessed at 3 months, 6 months, 9 months, and 12 months' post-fracture.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - CBT (Experimental): Participants in this arm will receive cognitive behavioural therapy (CBT). Participants will complete a series of online modules via a mobile application in addition to standard of care for their fracture injury. Participants will be assigned a dedicated CBT therapist, and receive feedback and support from their therapist via in-app messaging. The CBT program will last approximately 6-8 weeks.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Control (No Intervention): Participants in the control arm of the study will receive standard of care treatment for their fracture(s) but will not receive any Cognitive Behavioral Therapy.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Participants who are randomized to the CBT intervention will be encouraged to begin CBT immediately following randomization. The CBT intervention will focus on addressing maladaptive beliefs related to pain and recovery as well as teaching skills to enhance coping and management of pain symptoms. The specific focus of CBT sessions will be informed by each individual patient's responses to baseline questionnaires. All other aspects of post-operative care will be at the discretion of participant's surgeon.
  Other Names: CBT
  Arms: Intervention - CBT

SUMMARY:
Psychological factors such as stress, distress, anxiety, depression, and poor coping strategies may be associated with ongoing pain following injuries such as fractures. To study this relationship, patients will undergo cognitive behavioural therapy (CBT) which is designed to modify such thoughts with the goal of reducing ongoing pain and improving quality of life. The goal of this study is to determine if CBT, versus usual care, reduces the prevalence of moderate to severe persistent post-surgical pain (PPSP) over 12-months post-fracture in patients with an open or closed fracture of the appendicular skeleton, treated with internal fixation.

DETAILED DESCRIPTION:
The relationship between psychological factors, behaviors, and cognitive processes and the sensation of pain is well documented. Stress, distress, anxiety, depression, catastrophizing, fear-avoidance behaviors, and poor coping strategies appear to have a significant positive relationship with both acute and chronic pain. Evidence suggests that these psychological factors can cause alterations along the spinal and supraspinal pain pathways which influence the perception of pain. Previous studies suggest that patients' beliefs and expectations may be associated with clinical outcomes, including self-reported pain. Previous studies in trauma patients have demonstrated patients' beliefs and expectations regarding their recovery following surgery are associated with functional limitations, lower rates of return to work, and reduced quality of life one year after injury. Furthermore, up to two thirds of patients with operative managed extremity fractures demonstrate unhelpful illness beliefs that increase risks of negative outcomes, including persistent pain. Psychological interventions, such as cognitive behavioural therapy (CBT), that are designed to modify unhelpful beliefs and behaviours have the potential to reduce persistent post-surgical pain and its associated effects among trauma patients.

Our primary objective is to determine if CBT, versus usual care, reduces the prevalence of moderate to severe PPSP over 12 months post-fracture in participants with an open or closed fracture of the appendicular skeleton. Our secondary objectives are to determine if CBT, versus usual care: 1) increases physical functioning, 2) improves mental functioning, 3) accelerates return to function, 4) reduces pain severity, and 5) reduces pain interference over 12 months post-fracture, and 6) reduces the proportion of participants prescribed opioid class medications at 6 and 12 months post-fracture. This trial is a multi-centre randomized controlled trial (RCT) of 1,000 participants with an open fracture of the appendicular skeleton or closed fracture of the lower extremity or pelvis treated with internal fixation.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 18 years and older.
* Presenting to fracture clinic within 2-12 weeks following an acute open or closed fracture of the appendicular skeleton. Patients with multiple fractures may be included.
* Fracture treated operatively with internal fixation.
* Willing to participate in CBT.
* Language skills and cognitive ability required to participate in CBT (in the judgement of site research personnel).
* Consistent access to a smart phone and/or tablet that is capable of running the CBT provider's application.
* Provision of informed consent.

Exclusion Criteria:

* Fragility fracture.
* Stress fracture.
* Concomitant injury which, in the opinion of the attending surgeon, is likely to impair function for as long as or longer than the patient's extremity fracture.
* Among patients who are fully weightbearing, those not experiencing any pain in the fracture region.
* Active psychosis.
* Active suicidality.
* Active substance use disorder that, in the judgement of the treating surgeon, would interfere in the patient's ability to partake in the CBT and/or the trial.
* Already participating in, or planning to, start other psychological treatments (including CBT) within the duration of the study (12 months).
* Anticipated problems, in the judgement of study personnel, with the patient participating in CBT intervention and/or returning for follow-up.
* Incarceration.
* Currently enrolled in a study that does not permit co-enrolment in other trials.
* Previously enrolled in the COPE trial.
* Other reason to exclude the patient, as approved by the Methods Centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1024 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
The prevalence of moderate to severe Persistent Post-Surgical Pain at 12 months' post-fracture | 12 months post-fracture
  The primary outcome is PPSP according to the World Health Organization's (WHO) proposed definition.
  The WHO's definition requires 4 criteria for the diagnosis of PPSP: 1) Pain that began after surgery or a tissue trauma is experienced; 2) The pain is in an area of preceding surgery or tissue trauma, 3) The pain persisted for at least three months after the initiating event, and 4) The pain is not better explained by an infection, a malignancy, a pre-existing pain condition or any other alternative cause.

SECONDARY OUTCOMES:
Short Form 36 (SF-36) | 12 months post-fracture
  General health related quality of life will be assessed by the SF-36. The SF-36 is an established, reliable and validated health status measure. It is a self-administered, 36-item questionnaire that measures health-related quality of life in 8 domains related to physical, social, mental, and emotional functioning, bodily pain, and general health. Both physical and mental summary scores can be obtained. Each domain is scored separately from 0 (lowest level) to 100 (highest level).
Return to Function Questionnaire | 12 months post-fracture
  Return to function will be measured by when participants' return to work, household activities, and leisure activities, as well as when they achieve 80% of their pre-injury function. The return to function outcome will be assessed using the Return to Function questionnaire.
Brief Pain Inventory-Short Form (BPI-SF) | 12 months post-fracture
  The Brief Pain Inventory (BPI) assess pain severity and its impact on function. Participants will rate their pain on a scale from 0-10 (0 being No Pain, and 10 being Pain as bad as you can imagine). Participants will also rate how pain has interfered with their every day life on a scale from 0-10 (0 being Does not interfere, and 10 being Completely Interferes).
Opioid Use | 12 months post-fracture
  Patient-reported use of opioid class medications. To determine if CBT versus usual care reduces the proportion of participants taking opioid class medications at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Sprague, PhD, Principal Investigator — McMaster University; Jason Busse, PhD, Principal Investigator — McMaster University
Locations (10):
- United States (6):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Maryland - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland - Capital Region Medical Center, Largo, Maryland
  - Beth Israel Deaconess Medical Centre, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Centre, Lebanon, New Hampshire
  - PRISMA Health, Greenwood, South Carolina
- Canada (4):
  - University of Calgary - Foothills Hospital, Calgary, Alberta
  - Memorial University Newfoundland, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario

REFERENCES:
- [Derived] Gouveia K, Sprague S, Gallant JL, MacRae S, Del Fabbro G, Bzovsky S, McKay P, Johal H, Busse JW; COPE Investigators. Cognitive Behavioural Therapy to Optimize Post-Operative Recovery (COPE): a randomized controlled feasibility trial in extremity fracture patients. Pilot Feasibility Stud. 2025 Jan 11;11(1):3. doi: 10.1186/s40814-024-01592-3. PMID 39799376
- [Derived] COPE Investigators. Cognitive Behavioural Therapy to Optimize Post-Operative Fracture Recovery (COPE): protocol for a randomized controlled trial. Trials. 2022 Oct 22;23(1):894. doi: 10.1186/s13063-022-06835-3. PMID 36273187

DOCUMENTS (6):
  • Statistical Analysis Plan: Version 1.0 (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_000.pdf
  • Statistical Analysis Plan: Version 2.0 (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_001.pdf
  • Statistical Analysis Plan: Version 3.0 (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_002.pdf
  • Statistical Analysis Plan: Version 4.0 (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_003.pdf
  • Statistical Analysis Plan: Version 5.0 (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_004.pdf
  • Statistical Analysis Plan: Version 5.0_Signed (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04274530/SAP_005.pdf